CLINICAL TRIAL: NCT02829840
Title: Phase I/II, Dose-Escalation Study of Ponatinib, a FLT3 Inhibitor, With and Without Combination of 5-Azacytidine, in Patients With FLT3-Mutated Acute Myeloid Leukemia (AML)
Brief Title: Dose-Escalation Study of Ponatinib, a FLT3 Inhibitor, With and Without Combination of 5-Azacytidine, in Patients With FLT3-Mutated Acute Myeloid Leukemia (AML)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1083; NCI-2016-01187 (Other: NCI CTRP)
Record Dates: First submitted 2016-07-05; First posted 2016-07-12 (Estimated); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Leukemia; FLT3-Mutated Acute Myeloid Leukemia; FLT3-Mutated High-Risk Myelodysplastic Syndrome
Keywords: Leukemia; FLT3-Mutated Acute Myeloid Leukemia; FLT3-Mutated High-Risk Myelodysplastic Syndrome; Acute Myeloid Leukemia; AML; Myelodysplastic Syndrome; MDS; Ponatinib; Iclusig; AP24534; 5-azacytidine; Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — ponatinib; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort #1 (Experimental): Cohort #1: Participants with no previous leukemia therapy (including no previous FLT3 inhibitor therapy) for either: a) front-line treatment of elderly (age 65 and greater) FLT3-mutated AML patients, or b) patients unable or unwilling to receive standard intensive therapy.
  Part 1: Ponatinib at starting dose of 30 mg by mouth every day for one 28 day cycle. If disease does not respond to ponatinib alone, participant continues on to Part 2 of study.
  Part 2 Phase I Dose Escalation: Ponatinib at starting dose of 30 mg by mouth every day of a 28 day cycle. 5-azacytidine at dose of 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) for on Days 1-7 of every 28 day cycle.
  Part 2 Phase II Dose Expansion: Ponatinib at maximum tolerated dose from Phase I by mouth every day of a 28 day cycle. 5-azacytidine 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) on Days 1-7 of every 28 day cycle.
  Interventions: Drug: Ponatinib; Drug: 5-azacytidine; Behavioral: Phone Calls
- Cohort #2 (Experimental): Cohort #2: Participants with relapsed/refractory FLT3-mutated AML that have not received prior FLT3 inhibitor therapy.
  Part 1: Participants receive Ponatinib at starting dose of 30 mg by mouth every day for one 28 day cycle. If disease does not respond to ponatinib alone, participant continues on to Part 2 of study.
  Part 2 Phase I Dose Escalation: Ponatinib at starting dose of 30 mg by mouth every day of a 28 day cycle. 5-azacytidine at dose of 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) for on Days 1-7 of every 28 day cycle.
  Part 2 Phase II Dose Expansion: Ponatinib at maximum tolerated dose from Phase I by mouth every day of a 28 day cycle. 5-azacytidine 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) on Days 1-7 of every 28 day cycle.
  Interventions: Drug: Ponatinib; Drug: 5-azacytidine; Behavioral: Phone Calls
- Cohort #3 (Experimental): Cohort #3: Participants with relapsed/refractory FLT3-mutated AML, that have received previous FLT3 inhibitor therapy (including, but not limited to, quizartinib, crenolanib, sorafenib, other FLT3 inhibitors).
  Part 1: Participants receive Ponatinib at starting dose of 30 mg by mouth every day for one 28 day cycle. If disease does not respond to ponatinib alone, participant will continue on to Part 2 of study.
  Part 2 Phase I Dose Escalation: Ponatinib at starting dose of 30 mg by mouth every day of a 28 day cycle. 5-azacytidine at dose of 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) for on Days 1-7 of every 28 day cycle.
  Part 2 Phase II Dose Expansion: Ponatinib at maximum tolerated dose from Phase I by mouth every day of a 28 day cycle. 5-azacytidine 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) on Days 1-7 of every 28 day cycle.
  Interventions: Drug: Ponatinib; Drug: 5-azacytidine; Behavioral: Phone Calls

INTERVENTIONS:
Drug: Ponatinib — Part 1: Ponatinib at starting dose of 30 mg by mouth every day for one 28 day cycle.
  Part 2 Phase I Dose Escalation: Ponatinib at starting dose of 30 mg by mouth every day of a 28 day cycle.
  Part 2 Phase II Dose Expansion: Ponatinib at maximum tolerated dose from Phase I by mouth every day of a 28 day cycle.
  Other Names: Iclusig; AP24534
Drug: 5-azacytidine — Part 2 Phase I Dose Escalation: 5-azacytidine at dose of 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) for on Days 1-7 of every 28 day cycle.
  Part 2 Phase II Dose Expansion: 5-azacytidine 75 mg/m2/d administered subcutaneously (SQ) or intravenously (IV) on Days 1-7 of every 28 day cycle.
  Other Names: Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Azacytidine
Behavioral: Phone Calls — About 30 days after end-of-study visit, study staff calls participant and asks if they have had any side effects and/or started any new treatment(s).
  If disease appears to be responding to study drugs, study staff calls participant every 3-6 months for up to 5 years and asks how they are doing and about any side effects they may be having.

SUMMARY:
The goal of Part 1 of this clinical research study is to learn if ponatinib alone can help to control FLT3-mutated AML or FLT3-mutated high-risk MDS. The safety of this drug will also be studied.

The goal of Part 2 of this clinical research study is to find the highest tolerable dose of ponatinib in combination with 5-azacytidine and to learn if the highest dose level found can help to control FLT3-mutated AML or FLT3-mutated high-risk MDS. The safety of this combination will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If participant is found to be eligible to take part in this study, they will be assigned to either Part 1 or Part 2 based on when they join this study.

If participant is enrolled in Part 1, they will receive ponatinib alone for the first cycle. If the doctor thinks it is needed, the dose level may be increased. If the disease does not respond to ponatinib alone, participant will continue on to Part 2 of this study.

Part 2 of this clinical research study will have 2 phases: Phase 1 (dose escalation) and Phase 2 (dose expansion).

In Part 2, participant will be assigned to a study group based on when they join this study. Up to 3 groups of 30 participants will be enrolled in Phase 1 of Part 2, and up to 60 participants will be enrolled in Phase 2.

If participant is enrolled in Phase 1, the dose of ponatinib they receive will depend on when they join this study. The first group of participants will receive the lowest dose level of ponatinib. Each new group will receive a higher dose of ponatinib than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of ponatinib is found.

If participant is enrolled in Phase 2, they will receive ponatinib at the highest dose that was tolerated in Phase 1.

All participants in Part 2 will receive the same dose level of 5-azacytidine.

Study Drug Administration:

Each study cycle is 28 days.

Participant will take ponatinib tablets by mouth 1 time every day while they are on study. Participant should swallow the tablets whole. Participant should not crush them.

If participant is enrolled in Part 2, they will receive 5-azacytidine either by vein over about 1 hour or as an injection under the skin on Days 1-7 of each study cycle or on Days 1-5, 8, and 9 of each study cycle (if the clinic is closed on a weekend).

If the doctor thinks it is needed, the dose level, dosing schedule, or study cycle may be changed and/or delayed. The study doctor will discuss any changes with participant.

Study Visits:

On Day 1 of each cycle (+/- 4 days), participant will have a physical exam.

On Day 1 (+/-1 day) of Cycles 1-3 and then every 3 cycles after that (Cycles 6, 9, 12, and so on), participant will have an EKG.

On Day 1 of Cycle 2 and then every 3 cycles after that, participant will have an ECHO or MUGA performed.

One (1) time each week during Cycles 1-3 and then 1 time every 2-4 weeks after that, blood (about 1 tablespoon) will be drawn for routine tests. Participant may be able to have these blood draws performed at a local lab or clinic that is closer to their home. The results of the testing will be sent to MD Anderson for review.

On Day 28 (+/- 7 days) of Cycles 1, 3, and then every 1-3 cycles after that, participant will have a bone marrow aspiration/biopsy to check the status of the disease.

One (1) time every 3 cycles, if participant can become pregnant, blood (about 1-2 tablespoons) will be drawn for a pregnancy test.

At any time while participant is on study, if the doctor thinks it is needed:

* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* Participant may have a bone marrow aspiration/biopsy to check the status of the disease.

Length of Study:

Participant will receive ponatinib alone or ponatinib and 5-azacytidine for as long as the doctor thinks it is in their best interest. Participant will no longer be able to take the study drugs if the disease gets worse, if intolerable side effects occur, or if they are unable to follow study directions.

Patient's participation on the study will be over after the follow-up visits.

End-of-Study Visit:

Within 14 days after participant's last dose of study drug(s):

* Participant will have a physical exam.
* Blood (about 2-3 tablespoons) will be drawn for routine tests.
* If the doctor thinks it is needed, participant will have a bone marrow aspirate/biopsy to check the status of the disease.

Follow-Up:

About 30 days after the end-of-study visit, a member of the study staff will call participant to ask if they have had any side effects and/or started any new treatment(s). This call should last about 5 minutes. If the study staff thinks it is needed, participant may also be asked to come into the clinic for a physical exam.

Long-Term Follow-Up:

If the disease appears to be responding to the study drugs, a member of the study staff will call participant every 3-6 months for up to 5 years to ask how they are doing and about any side effects they may be having. Each call should last about 5 minutes. Participant may also be asked to come into the clinic for a physical exam, if the study staff thinks it is needed.

This is an investigational study. 5-azacytidine is FDA approved and commercially available for the treatment of myelodysplastic syndrome (MDS). Ponatinib is commercially available and FDA approved for the treatment of specific groups of chronic myeloid leukemia (CML) participants. Their use in this study is considered investigational. The study doctor can explain how the study drugs are designed to work.

Up to 132 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients should have a diagnosis of AML (de novo or transformed from hematologic malignancies), MDS or chronic myelomonocytic leukemia (CMML) with one of the following features: (A) Patients with MDS or CMML should have failed prior therapy with a hypomethylating agent and/or with lenalidomide (Cohorts 2 and 3). (B) Patients with AML should have failed any prior therapy or have relapsed after prior therapy (Cohorts 2 and 3). For patients in Cohort 3 prior therapy should have included a FLT3 inhibitor. (C) Patients with MDS or CMML who received therapy with a hypomethylating agent and progress to AML are eligible at the time of diagnosis of AML regardless any prior therapy for AML. The World Health Organization (WHO) classification will be used for AML. These patients will be assigned to Cohort 1. Patients with MDS, CMML or AML who have received no prior therapy are eligible if age 65 and greater or if, at the time of enrollment, are not candidates to receive or refuse standard therapy (Cohort 1 only)
2. Patients should have a FLT3 mutation, either ITD or kinase domain mutation or activation loop mutation.
3. Age >/= 18 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Status </= 2
5. Adequate hepatic (serum total bilirubin < 2.0 x upper limit normal (ULN) (or < 3.0 x ULN if deemed to be elevated due to leukemia or Gilbert's syndrome), alanine aminotransferase and/or aspartate transaminase < 3.0 x ULN (or < 5.0 x ULN if deemed to be elevated due to leukemia), and renal function (creatinine 2x ULN or glomerular filtration rate (GFR) > 50) function.
6. Left ventricular ejection fraction (LVEF) at least 40% by multiple gated acquisition (MUGA) scan or echocardiogram (ECHO)
7. Patients must provide written informed consent.
8. In the absence of rapidly progressing disease, the interval from prior treatment to time of initiation of ponatinib administration will be at least 2 weeks for cytotoxic agents OR at least 5 half-lives for cytotoxic/non-cytotoxic agents. Use of one dose of cytarabine (up to 2 g/m2) or hydroxyurea for patients with rapidly proliferative disease is allowed before the start of study therapy and for the first eight weeks on study therapy from the day of enrollment, either prior to or concomitantly with ponatinib administration initially to control the peripheral blast count. Concurrent therapy for central nervous system (CNS) prophylaxis or continuation of therapy for controlled CNS disease is permitted. Controlled CNS leukemia is defined by the absence of active clinical signs of CNS disease and no evidence of CNS leukemia on the most recent 2 simultaneous cerebrospinal fluid (CSF) evaluations.
9. Women of childbearing potential must practice contraception. Females of childbearing potential: Recommendation is for 2 effective contraceptive methods during the study. Adequate forms of contraception are double barrier methods (condoms with spermicidal jelly or foam and diaphragm with spermicidal jelly or foam), oral, depo provera, or injectable contraceptives, intrauterine devices, and tubal ligation. Male patients with female partners who are of childbearing potential: Recommendation is for male and partner to use at least 2 effective contraceptive methods, as described above, during the study.
10. Females must be surgically or biologically sterile or postmenopausal (amenorrheic for at least 12 months) or if of childbearing potential, must have a negative urine pregnancy test within 72 hours or serum pregnancy test within 2 weeks of signing the Informed Consent document.
11. Women of childbearing potential must agree to use an adequate method of contraception during the study and until 3 months after the last treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study until 3 months after the last treatment. Adequate methods of contraception include: (A) Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception. (B) Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
12. 11 (Cont'd): (C) Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient (D) Combination of any of the two following (a+b or a+c or b+c): (1) Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception (B) Placement of an intrauterine device (IUD) or intrauterine system (IUS). (C) Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository In case of use of oral contraception, women should have been stable on the same pill before taking study treatment. Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction.
13. 11 (Cont'd) Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
14. 1 (Cont'd) not considered candidates for intensive remission induction chemotherapy at time of enrollment based on EITHER: 1. >/= 75 years of age OR 2. <75 years of age with at least 1 of the following: A. Poor performance status (ECOG) score of 2-3 B. Clinically significant heart or lung comorbidities, as reflected by at least 1 of: (i) Left ventricular ejection fraction </= 50%, (ii) Lung diffusing capacity for carbon monoxide (DLCO) </= 65% of expected, (iii) forced expiratory volume in 1 second (FEV1) </= 65% of expected, (iv) congestive heart failure (CHF) C. Serum creatinine >2 mg/dL, are on dialysis or have history of renal transplant. D. Other contraindication(s) to anthracycline therapy (must be documented). E. Other comorbidity the investigator judges incompatible with intensive remission induction chemotherapy, which must be documented and approved by the PI before randomization.

Exclusion Criteria:

1. Patients with known allergy or hypersensitivity to ponatinib, or 5-azacytidine, or any of their components.
2. Patients who have received any treatment of ponatinib prior to study entry.
3. History of acute pancreatitis within 1 year of study or history of chronic pancreatitis.
4. History of alcohol abuse.
5. Uncontrolled infection at the time of enrollment. Infections controlled on concurrent anti-microbial agents are acceptable, and anti-microbial prophylaxis per institutional guidelines is acceptable.
6. Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year.
7. Cardiac Symptoms: Patients meeting the following criteria are not eligible: History of unstable angina, myocardial infarction, transient ischemic attack (TIA), stroke, peripheral arterial occlusive disease, venous thromboembolism or pulmonary embolism. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes). Prolonged corrected QT interval (QTc) interval on pre-entry electrocardiogram (> 470 msec) on both the Fridericia and Bazett's correction. Symptomatic congestive heart failure within 3 months prior to first dose of ponatinib (NYHA class III or IV).
8. Patients with uncontrolled hypertension (defined as sustained stage 2 hypertension, i.e., systolic BP >/=160 mmHg or diastolic BP >/=100 mmHg) with or without medical therapy.
9. Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes (unless these can be changed to acceptable alternatives).
10. Taking any medications or herbal supplements that are known to be strong inhibitors of CYP3A4 within at least 14 days before the first dose of ponatinib.
11. Patients who have had any major surgical procedure within 14 days of Day 1.
12. Patients unwilling or unable to comply with the protocol.
13. History of significant bleeding disorder unrelated to cancer, including: • Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease) • Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
14. Patients with inflammatory or chronic functional bowel disorder, such as Crohn disease, inflammatory bowel disease, or gastrointestinal graft versus host disease that in the opinion of the investigator may interfere with absorption of ponatinib or increase the risk of serious complications.
15. Any other medical, psychological, or social condition that may interfere with study participation or compliance, or compromise patient safety in the opinion of the investigator.
16. Known active hepatitis B virus (HBV) or C virus (HCV) infection; or known to be positive for HCV ribonucleic acid (RNA) or HBsAg (HBV surface antigen).
17. Known human immunodeficiency virus (HIV) infection.
18. Patients who at the time of enrollment, are willing and eligible to receive a stem cell transplant will not be eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Ponatinib | 28 days
  MTD defined as highest dose level with </= 1 out of 6 patients experience a dose limiting toxicity (DLT) during the first 28 days of treatment. DLT defined as clinically significant non-hematologic adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications.
Rate of Composite Complete Remission (CRc) | 84 days
  CRc defined as complete remission (CR), complete remission with incomplete platelet recovery (CRp), or complete remission with incomplete blood count recovery (CRi). Response defined by achievement of CRc at any point in time within the first 3 cycles of therapy, or prior to going off study, for those patients discontinuing treatment before completion of 3 cycles of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org